CLINICAL TRIAL: NCT06796101
Title: The Effect of Auricular Vagus Nerve Stimulation and Controlled Breathing Exercises on Performance and Autonomic Nervous System in Healthy Individuals
Brief Title: The Effect of Auricular Vagus Nerve Stimulation and Controlled Breathing Exercises on Performance and Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Okan Sahin, Principal Investigator, PT (Physiotherapist), MSc, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ODRP-2025
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Health People; Physical Activity; Autonomic Nerveus System; Vagus Nerve Stimulations
Keywords: Transcutaneous vagus nerve stimulation; Performance; Controlled breathing exercises; Autonomic nervous system; recreactional
MeSH Terms: conditions — Motor Activity | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Individuals who are moderately physically active according to the physical activity scale between the ages of 18-35 who met the inclusion criteria will be included in the study. The sample size of the study is calculated as 64 and randomized to vagus stimulation and controlled breathing exercise groups. All evaluations of the participants will be held at Bahçeşehir University Faculty of Health Sciences Biomechanics chiropractic laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneus vagus nerve stimulation (Experimental): This group will receive Transcutaneous vagus nerve stimulation from bilateral ear for two weeks, 10 sessions.
  Interventions: Device: Vagus Nerve Stimulation
- Controlled breathing exercise group (Experimental): Controlled breathing exercises include thoracic expansion exercises, Nadi Shodhana Pranayama, Bhramari Pranayama, Kapalabhati and Physiological-sighing exercises.
  Interventions: Other: Controlled breathing exercises

INTERVENTIONS:
Device: Vagus Nerve Stimulation — In the study, CE certified vagus nerve stimulation device Vagustim will be used. Transcutaneous auricular vagus nerve stimulation will be applied bilaterally. The stimulation pulse width is 300 microseconds, frequency is 10 Hz and will be applied biphasically for 20 minutes.
  Arms: Transcutaneus vagus nerve stimulation
Other: Controlled breathing exercises — A controlled breathing exercise group will continue for a total of 2 weeks and will receive 10 sessions of 20 minutes per day.
  The thoracic expansion exercise will be performed in 10 repetitions. In each intervention session, 2 sets of nadi shodhana pranayama consisting of 8 respiratory cycles will be applied to the patients, with a 2-minute rest period between the sets. Kapalabhati will be practised for 3 minutes, with 15 quick breaths in 10 seconds followed by a 20-second break (a total of 30 breaths per minute). In each session, 2 sets of bhramari pranayama consisting of 10 breathing cycles will be performed at a low respiratory rate, with a 1-minute rest period between sets. The physiological sigh exercise involves the first inspiration phase being 1 second, the second phase 0.25 seconds, and the exhalation 2 seconds for 3 minutes.
  Arms: Controlled breathing exercise group

SUMMARY:
There are many studies in the literature on transcutaneous vagus nerve stimulation (VNS) and controlled breathing exercises (CBE), but there are limited studies examining the effects of both interventions on performance and the autonomic nervous system.

The investigators aim to contribute to the literature by examining the effects of VNS and CBE on performance and the autonomic nervous system in moderately physically active individuals and their superiority over each other.

DETAILED DESCRIPTION:
The sympathetic and parasympathetic divisions of the autonomic nervous system affect the function of many organs, glands, and involuntary muscles in the body. The sympathetic and parasympathetic nervous systems often play opposing roles in the body, one is suppressed when the other increases activity. With the beginning of exercise or sports activity, sympathetic activity in the body increases and after a certain period reaches a plateau value at maximum activity. With the end of sports activity, the suppressed parasympathetic activity increases, and the sympathetic system returns to its resting state over time.

Low sympathetic activity and/or high parasympathetic activity and low heart rate before training or exercise can be considered as performance indicators. It also indicates that recovery from the previous training or exercise is adequate. Parasympathetic system activation continues for up to 48 hours after exercise. If the exercise is intense and persistent, parasympathetic system activity can last up to 72 hours. In addition, due to the increase in anaerobic respiratory rate during exercise, there may be decreases in parasympathetic reactivation.

Transcutaneous vagus nerve stimulation (VNS) can affect cardiovascular parameters both at rest and during exercise. VNS improves autonomic modulation and positively reduces pain and fatigue associated with cycling exercise. On the other hand, VNS is particularly useful in reducing pain and fatigue during and after competition.

Slow breathing modulates the activity of the vagus nerve. Controlled breathing exercises (CBE) directly affect the respiratory rate, which can lead to faster physiological and psychological calming effects by increasing vagal tone during slow expiration. CBE increase heart rate variability in healthy participants.

The investigators aim to contribute to the literature by examining the effects of VNS and CBE on performance and the autonomic nervous system in moderately physically active individuals and their superiority over each other.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a moderate level of physical activity according to the International Physical Activity Scale
* No orthopedic obstacle to exertion
* Being male

Exclusion Criteria:

* Having any active or chronic disease
* Having cooperation problems
* Using regular medication for any chronic condition within the last year
* Being a smoker
* Having had heart surgery
* Having had surgery on the respiratory system

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Performance | Baseline and 2 weeks.
  Individuals will be taken to the treadmill and the distance and time taken until the maximum heart rate value reaches 80% will be recorded. The maximum heart rate value will be determined for each individual according to the formula 220-age.
  The participants will walk at a speed of 2 km/h for 1 minute, at a speed of 4 km/h for 1 minute and at a speed of 6 km/h, and the distance and time taken until the maximum heart rate reaches 80% will be recorded. In the termination phase of the run, a walk will be performed at a speed of 4 km/h for 1 minute and a speed of 2 km/h for 1 minute and will be completed.
Autonomic nervous system | Baseline and 2 weeks.
  Heart rate change will be evaluated for the evaluation of the autonomic nervous system. Polar H9 heart rate sensor chest strap and wristwatch will be used to measure analytical heart rate change. During the assessment, the participant will be seated in a chair and the Polar system chest strap will be placed just above the sternum, and ultrasound gel will be used to increase the sensor's conductivity. This method is valid with an electrocardiogram. Heart rate variability parameters such as RMSSD, LF, and HF will be measured.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline
  International Physical Activity Questionnaire is used to determine the activity levels of individuals. IPAQ Short Form, consisting of seven questions, provides information on the time spent walking, moderate-intensity and vigorous-intensity activities, and the time spent sitting. The calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.
Modified Borg Scale | Baseline and 2 weeks.
  Developed by Gunnar Borg, this scale includes values from 1 to 10 and difficulty statements written next to some of these values. This scale, used to determine the intensity of exercises and training, is a subjective method in which individuals determine the difficulty level of the exercise and training themselves.
Perceived Stress Scale | Baseline and 2 weeks.
  It is used to determine the stress level of individuals. The scale consists of 10 items in total. The items of the scale are answered using a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score varies between 0-40. It is concluded that as the score obtained from the scale increases, the perceived stress increases.
Blood Pressure Measurement | Baseline and 2 weeks.
  Blood pressure measurement will be done using an Omron brand digital wrist type blood pressure monitor. Before taking the measurement, individuals will be asked to rest for at least 5 minutes to ensure that they are relaxed for accurate measurement.
Pulse | Baseline and 2 weeks.
  Pulse measurement will be done with a finger-type Pulse oximeter device.
Oxygen Saturation | Baseline and 2 weeks.
  Pulse oximetry is a noninvasive, painless and reliable method used to measure oxygen saturation (SpO2) in arterial blood. Oxygen saturation measurement will be done with a finger-type pulse oximetry device.

CONTACTS AND LOCATIONS:
Overall Officials: Okan ŞAHİN, PT, MSc, Principal Investigator — Bahçeşehir University; Ali Veysel ÖZDEN, MD, PHD, Study Director — Bahçeşehir University
Locations (1):
- Bahçesehir University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No